CLINICAL TRIAL: NCT05127629
Title: Comparison of Clinical Outcomes of Different Wound Closure Methods in Immediate Implant Placement in the Aesthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210205.V1
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Tooth Fracture; Tooth Decay
Keywords: Immediate implant placement
MeSH Terms: conditions — Tooth Fractures; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Procedure: Immediate implant placement; Procedure: Guided bone regeneration; Procedure: Wound closure with gelatin sponge
- Collagen matrix (Experimental)
  Interventions: Procedure: Immediate implant placement; Procedure: Guided bone regeneration; Procedure: Wound closure with collagen matrix

INTERVENTIONS:
Procedure: Immediate implant placement — After tooth extraction, a dental implant is placed immediately.
Procedure: Guided bone regeneration — After implant placement, the gap between implant and the buccal bone wall is filled with Bio-oss collagen.
Procedure: Wound closure with gelatin sponge — After guided bone regeneration, patient in the control group receive gelatin sponge for wound closure.
  Arms: Control
Procedure: Wound closure with collagen matrix — After guided bone regeneration, patient in the control group receive collagen matrix (Mucograft Seal) for wound closure.
  Arms: Collagen matrix

SUMMARY:
Implant-supported restorations have become one of the best treatment options for patients with tooth loss, with predictable long-term success rates and clinical outcomes. Immediate implant placement means the implant is placed immediately after tooth extraction. It can significantly reduce treatment time because extraction socket healing and implant osseointegration occur simultaneously. Immediate implant placement has many benefits, reducing the overall treatment time, reducing the patient's surgical procedures, and reducing surgical trauma (no flap reversal). However, the treatment also has significant limitations, including the inability to predict the possibility of bone and soft tissue healing, and the possibility of subsequent unfavorable esthetic outcomes. However, the evidence regarding soft and hard tissue and aesthetic outcomes in patients treated with immediate implants in the aesthetic area remains inconclusive. As the aesthetic success of implant restorations is increasingly valued over implant survival, there are significant clinical benefits to addressing immediate implant bone tissue resorption and soft tissue deficiencies and improving the aesthetic outcome of immediate implant restorations.

To address the potential health and aesthetic problems associated with soft and hard tissue deficiencies around dental implants, bone grafting in the jumping gap and soft tissue grafting procedures are often performed. According to literature, autologous soft tissue grafts have shown the best clinical and histological results in soft tissue regeneration techniques. However, it requires removal of tissue from the patient's donor area, which can add additional trauma. In contrast, gelatin sponges, currently commonly used as wound closure materials, are only hemostatic and rapidly absorbed postoperatively, and do not provide protection of hard and soft tissue augmentation. Collagen matrix has recently been introduced for keratinized gingival augmentation and has shown encouraging results in preclinical and clinical studies, but more information is needed to confirm its clinical efficacy. Mucograft® Seal is a porcine collagen matrix with a bilayer structure, a dense and slowly absorbing layer and a spongy layer that stabilizes blood clots and allows soft tissue cells to penetrate. Human gingival fibroblasts cultured on Mucograft® were demonstrated to have good proliferative properties and cell viability as scaffold material. In dog extraction sites, preliminary results suggest that the combination of Mucograft® and Bio-Oss Collagen may be an effective method for alveolar ridge preservation. Mucograft® Seal can be used in combination with Bio-Oss Collagen® for alveolar ridge preservation after tooth extraction.

The research hypothesis is that the use of a collagen matrix to seal the wound in immediate implant placement in aesthetic area will reduce buccal bone resorption and increase the width and thickness of the soft tissue at the implant site.

Therefore, we designed this comparative clinical trial in which patients accept immediate implant placement in aesthetic area. The implant is placed after tooth extraction, and bone graft material Bio-Oss Collagen® is placed in the jump gap, and the wound was closed by different means (collagen matrix or gelatin sponge randomly). The clinical examination, CBCT imaging and histological evaluations were performed to compare the differences in clinical efficacy of the two wound closure methods. The primary outcome is the buccal bone thickness change at the immediate implant site 4 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are at least 18 years old and in good health;
2. Single tooth in the maxillary anterior aesthetic area to be extracted for immediate implant placement;
3. The labial bone plate is intact and there is sufficient bone in the apical region to ensure initial stability.
4. Healthy intraoral soft tissues and no infection.

Exclusion Criteria:

1. Need to place more than 1 implant in the aesthetic area.
2. Heavy smokers (> 10 cigarettes/day).
3. Patients with physical diseases such as: uncontrolled diabetes (fasting glucose > 7.2 mmol/L, glycosylated hemoglobin > 7%), current intake of bisphosphonate medication, history of head and neck malignancy, history of head and neck radiotherapy, pregnancy or preparation for pregnancy, etc.
4. Patients with uncontrolled periodontitis and unstable periodontal status.
5. Lateral labial bone plate defect;
6. Missing teeth;
7. Allergic to titanium;

e. Those who do not wish to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Thickness of the buccal bone | 4 months after implant surgery
  Change in labial alveolar bone thickness, including alveolar bone thickness and implant bone powder thickness

SECONDARY OUTCOMES:
gingival thickness | 4 months after implant surgery
  Change of gingival thickness
success rate | 4 months after implant surgery
  success rate of implant
Wound healing | 2weeks and 4 months after implant surgery
  Wound healing status

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Implantology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
ngc